CLINICAL TRIAL: NCT03097224
Title: Prehabilitation Before Surgery in Colorectal Cancer With Improved Fast Track Rehabilitation : Part 2
Brief Title: Prehabilitation in Frail Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Caty Gilles, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Part 2
Record Dates: First submitted 2017-03-17; First posted 2017-03-31 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Colon Cancer; Fragility
MeSH Terms: conditions — Colonic Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): Tele-supervised prehabilitation
  Interventions: Behavioral: Prehabilitation
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Prehabilitation — Four weeks of tele-supervised prehabilitation
  Arms: Prehabilitation group

SUMMARY:
Objectives To investigate the impact of tele-supervised prehabilitation on functional capacity in frail colon cancer patients undergoing colorectal resection and to evaluate the effects of prehabilitation on muscle strength and endurance, quality of life (QoL), executive functions, fatigue and inflammatory and metabolic parameters.

Methods A randomized controlled trial will be conducted. Patients will be randomised into either a prehabilitation group (PREHAB) or a control group. Prehabilitation group will participate in a 4-week telerehabilitation before surgery while the control group will receive usual care and World Health Organization recommendations on physical activity for health before surgery. Program exercise will consist of three moderate-intensity aerobic and resistance sessions per week. Subjects will have assessments at baseline, pre-intervention and 8 weeks after surgery. The primary outcome will be functional capacity measured by using the 6-min walk test. The secondary outcomes will be: physical measurements, QoL, level of physical activity, executive functions, fatigue, body composition, blood test, energy expenditure.

DETAILED DESCRIPTION:
Objectives Primary objective: To assess if a 4-week tele-supervised prehabilitation is effective in improving post-operative cardio-respiratory fitness in frail colon cancer patients.

Secondary objectives : To examine if a 4-week preoperative tele-supervised prehabilitation has beneficial effects on muscle strength and endurance, on quality of life, on executive functions, on fatigue, on inflammatory parameters and on metabolic disruption pre-surgery.

Background In Belgium, colon cancer is the third most common cancer in men and the second most common in women and is the second cause of cancer death. Surgery is currently the primary treatment for stage I to III. Studies have shown that patients with poor preoperative physical fitness are less able to cope with the adverse effects of surgery and hospitalization resulting in increased risk of mortality, postoperative complications and functional recovery time. Moreover, approximately 60% of colon cancer patients are older than 70 years at diagnosis and more than 50% of older cancer patients have frailty or pre-frailty. Frailty is a state of vulnerability decreased functional reserve, impairment or dysregulation in several physiological systems, and reduced capacity to recover physiological homeostasis after a stress. Nowadays, no frail definition is clearly defined. One widely accepted definition uses the Fried criteria including the assessment of weight loss, physical exhaustion, physical activity level, grip strength and walking speed. Preoperative frail colon cancer patients have a significantly higher risk of adverse postoperative outcomes including institutionalization, length of stay, morbidity and mortality. It seems relevant to intervene during the preoperative period to improve the patient's functional capacity before the surgery, via physical training to overcome the stress of the surgery and to improve postoperative recovery. This process is called "prehabilitation". Structured and supervised programs have shown to be effective and feasible. However, time, resources and expensive care are often a barrier for the patient. Thereby, a home-based tele-supervising rehabilitation would be an attractive therapeutic option to offer a distinct advantage in this regard. To date, no study has studied the effects of tele-supervised prehabilitation in these "frail" patients.

Study design A single-blind, randomized, controlled trial will be conducted. Participants will be randomized into either a prehabilitation group or a control group. An assessor who will be blinded to group allocation will collect outcomes measures for each participant.

Study sample To be eligible for this study participants will need to meet the following criteria: diagnosis of colon cancer requiring surgery; more than 65 years of age; able to read, write and understand French; Frailty phenotype criteria ≥ 3. Frailty was assessed using the components of the Frailty Phenotype, which was first developed by Fried et al., which consists of five criteria: weight loss, exhaustion, low physical activity, slowness, and weakness.

Participants will be excluded if they have a physical impairment that would seriously impair physical mobility; the surgery is an emergency; have a neuropsychiatric disease.

Intervention Participants allocated to the prehabilitation group will undertake a telerehabilitation program that will start 4 weeks before the surgery while participants in the control group will receive usual care and World Health Organization recommendations on physical activity for health before surgery.

The telerehabilitation program will combine aerobic and resistance training three sessions per week. Each 60-min session will begin and end with a five-minute warm-up/cool. The warm-up will be followed by 25 minutes of aerobic training. Aerobic exercise can include brisk walking, jogging, cycling, or swimming according to patient's preference. The intensity of the exercise was set between 60 à 75% of maximum heart rate (maximal heart rate=220 - age). And between 12 and 16 on Borg's Rating of Perceived Exertion Scale. Each participant will wear a heart monitor. The aerobic training will be followed by resistance exercise performed on eight exercises targeting major muscle groups (abdominal, hamstring, quadriceps, triceps, gluteus maximus, paraspinal muscles and shoulder muscles). Intensity must be between 12 and 16 on the Borg's Rating of Perceived Exertion Scale. A physiotherapist will provide detailed information about the program. The patient will receive a brochure in which there will be descriptions and pictures of exercises and a video including the resistance program was recorded on a website. The researcher will conduct weekly telephone calls with the participants. The aim of these calls will be to solve any problems of carrying out the training sessions and to discuss about possible adverse events. Moreover, the researcher will give messages of support and encouragement to improve adherence to the program.

Outcome measures Outcome measures will be assessed at three time points: at baseline (T0), one day before the scheduled date of surgery (T1) and 8 weeks after the surgery (T2).

Primary outcome will be cardiorespiratory fitness 6min walk test). Secondary outcomes will be muscle strength and endurance (isokinetic dynamometer and 1-min sit-to-stand-test), quality of life (EQ-5D-3L questionnaire); level of physical activity (International Physical Activity Questionnaire Short Form); fatigue (Functional Assessment of Cancer Therapy: Fatigue); executive functions (Trail Making test and fluency verbal test) ; blood test (neutrophil lymphocyte ratio, C reactive protein, fasting glucose, fasting insulin and cholesterol will be measured by bioelectrical impedance analysis); energy expenditure (Sensewear® armband).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colon cancer requiring surgery
* More than 65 years of age;
* Able to read, write and understand French;
* Frailty phenotype criteria ≥ 3

Exclusion Criteria:

* The participants have a physical impairment that would seriously impair physical mobility;
* the surgery is an emergency;
* The participants have a neuropsychiatric disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Cardiorespiratory is measured by a 6-minute walk test

SECONDARY OUTCOMES:
Change in muscle strength | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Muscle strength is measured by using an isokinetic dynamometer
Change in muscle endurance | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Muscle endurance is measured by using the "1-minute sit-to-stand-test" (number of sit-to-stand cycles during 1 minute)
Change in quality of life | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Quality of life is measured by using the EQ-5D-3L questionnaire
Change in fatigue | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Fatigue is measured by using the Functional Assessment of Cancer Therapy: Fatigue questionnaire
Change in level of physical activity | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Level of physical activity is measured by using the International Physical Activity Questionnaire Short Form
Change in executive functions | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Executive functions is measured by using the Trail Making test
Change in executive functions | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Executive functions is measured by using the Fluency verbal test
Change in weight | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Weight (kg) is measured by using a bioelectrical impedance analysis
Change in lean body mass | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Lean body mass (kg) is measured by using a bioelectrical impedance analysis
Change in fat body mass | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Fat body mass (kg) is measured by using a bioelectrical impedance analysis
Energy expenditure | During 7 days before the surgery and during 7 days after the surgery
  Energy expenditure is measured by using the Sensewear® Armband
Change in Fasting glucose | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Fasting glucose is measured by a blood test
Change in Fasting insulin | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Fasting insulin is measured by a blood test
Change in cholesterol | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Cholesterol is measured by a blood test
Change in neutrophil/lymphocyte | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  Neutrophil/lymphocyte is measured by a blood test
Change in C-reactive protein | Assessments at baseline, one day before the surgery and 8 weeks after the surgery
  C-reactive protein is measured by a blood test
Adherence | Weekly through the intervention (during four weeks)
  Percentage of sessions completed

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Woluwé-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boereboom C, Doleman B, Lund JN, Williams JP. Systematic review of pre-operative exercise in colorectal cancer patients. Tech Coloproctol. 2016 Feb;20(2):81-9. doi: 10.1007/s10151-015-1407-1. Epub 2015 Nov 27. PMID 26614304
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Pallis AG, Papamichael D, Audisio R, Peeters M, Folprecht G, Lacombe D, Van Cutsem E. EORTC Elderly Task Force experts' opinion for the treatment of colon cancer in older patients. Cancer Treat Rev. 2010 Feb;36(1):83-90. doi: 10.1016/j.ctrv.2009.10.008. Epub 2009 Nov 26. PMID 19944536
- [Background] Lawrence VA, Hazuda HP, Cornell JE, Pederson T, Bradshaw PT, Mulrow CD, Page CP. Functional independence after major abdominal surgery in the elderly. J Am Coll Surg. 2004 Nov;199(5):762-72. doi: 10.1016/j.jamcollsurg.2004.05.280. PMID 15501119
- [Background] Wilson RJ, Davies S, Yates D, Redman J, Stone M. Impaired functional capacity is associated with all-cause mortality after major elective intra-abdominal surgery. Br J Anaesth. 2010 Sep;105(3):297-303. doi: 10.1093/bja/aeq128. Epub 2010 Jun 23. PMID 20573634
- [Background] Robinson TN, Wu DS, Pointer L, Dunn CL, Cleveland JC Jr, Moss M. Simple frailty score predicts postoperative complications across surgical specialties. Am J Surg. 2013 Oct;206(4):544-50. doi: 10.1016/j.amjsurg.2013.03.012. Epub 2013 Jul 20. PMID 23880071
- [Background] Millan M, Merino S, Caro A, Feliu F, Escuder J, Francesch T. Treatment of colorectal cancer in the elderly. World J Gastrointest Oncol. 2015 Oct 15;7(10):204-20. doi: 10.4251/wjgo.v7.i10.204. PMID 26483875
- [Background] Handforth C, Clegg A, Young C, Simpkins S, Seymour MT, Selby PJ, Young J. The prevalence and outcomes of frailty in older cancer patients: a systematic review. Ann Oncol. 2015 Jun;26(6):1091-1101. doi: 10.1093/annonc/mdu540. Epub 2014 Nov 17. PMID 25403592
- [Background] Chen X, Mao G, Leng SX. Frailty syndrome: an overview. Clin Interv Aging. 2014 Mar 19;9:433-41. doi: 10.2147/CIA.S45300. eCollection 2014. PMID 24672230
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Fagard K, Leonard S, Deschodt M, Devriendt E, Wolthuis A, Prenen H, Flamaing J, Milisen K, Wildiers H, Kenis C. The impact of frailty on postoperative outcomes in individuals aged 65 and over undergoing elective surgery for colorectal cancer: A systematic review. J Geriatr Oncol. 2016 Nov;7(6):479-491. doi: 10.1016/j.jgo.2016.06.001. Epub 2016 Jun 21. PMID 27338516
- [Background] Debes C, Aissou M, Beaussier M. [Prehabilitation. Preparing patients for surgery to improve functional recovery and reduce postoperative morbidity]. Ann Fr Anesth Reanim. 2014 Jan;33(1):33-40. doi: 10.1016/j.annfar.2013.12.012. Epub 2014 Jan 17. French. PMID 24440732
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub3. PMID 37162250
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252